CLINICAL TRIAL: NCT04708496
Title: Optimizing Malaria Treatment for HIV-Malaria Co-Infected Individuals by Addressing Drug Interactions Between Artemether-Lumefantrine and Efavirenz; a Randomized Controlled Trial
Brief Title: Optimizing Malaria Treatment for HIV-Malaria Co-infected Individuals
Acronym: OPTIMAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PK25
Record Dates: First submitted 2020-11-12; First posted 2021-01-14 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-01

CONDITIONS: HIV Coinfection; Malaria
MeSH Terms: conditions — HIV Infections; Malaria | interventions — Artemether, Lumefantrine Drug Combination; efavirenz; dolutegravir

STUDY DESIGN:
Intervention Model Description: A three arm single blind randomized trial. Study participants will be randomized to one of the 3 arms. Standard dose, double dose or 5 day course of Artemether-lumefantrine
Who Masked: Investigator
Masking Description: study physicians and laboratory technicians will be blinded to treatment group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard dose of Artemether lumefantrine (Experimental): Dose comparison-concurrent control In this arm, Participants receiving Efavirenz400mg based ART will be randomized to standard dose Artemether Lumefantrine when treating uncomplicated malaria in HIV-malaria co-infected participants
  Interventions: Drug: Artemether-lumefantrine
- Double dose Artemether lumefantrine (Experimental): Dose comparison concurrent control In this arm, Participants receiving Efavirenz based ART will be randomized to double dose Artemether Lumefantrine when treating uncomplicated malaria in HIV-malaria co-infected participants
  Interventions: Drug: Artemether-lumefantrine
- 5 day course of Artemether lumefantrine (Experimental): Dose comparison concurrent control In this arm, Participants receiving Efavirenz based ART will be randomized to 5 day course of Artemether Lumefantrine as opposed to the standard 3day course when treating uncomplicated malaria in HIV-malaria co-infected participants
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artemether-lumefantrine — A three-arm single blind Randomized Clinical Trial in which HIV-malaria co-infected individuals with uncomplicated malaria receiving efavirenz-based ART will be randomized to one of three arms; a standard dose of artemether-lumefantrine, or a double dose of artemether-lumefantrine, or a 5-day course of artemether-lumefantrine for treatment of uncomplicated malaria. Participants will be followed up for 42 days to determine safety, drug pharmacokinetics and malaria treatment outcomes.
  The 4th objective focuses on the interaction between Dolutegravir and Artemether Lumefantrine hence this will be a single blind pharmacokinetic trial among HIV-malaria co-infected individuals receiving Dolutegravir based ART and standard dose of artemether-lumefantrine for treatment of uncomplicated malaria.
  Other Names: Efavirenz; Dolutegravir

SUMMARY:
Optimal is a Randomized clinical trial to optimize treatment of malaria in HIV -malaria co infected patients. It has been demonstrated that, when the antimalarial drug Artemether Lumefantrine is co administered with Efavirenz based ART in HIV-malaria co-infected individuals, sub therapeutic levels of the drug are achieved hence resulting in poor malaria treatment outcomes.

The study then hypothesizes that, : HIV-malaria co-infected individuals receiving efavirenz-based ART plus a double-dose or 5-day course of artemether-lumefantrine will achieve higher and adequate artemether-lumefantrine serum concentrations with adequate 42-day treatment outcomes compared to individuals with HIV-malaria co-infection receiving efavirenz-based ART plus a standard-dose of artemether-lumefantrine.

DETAILED DESCRIPTION:
Malaria and HIV have significant interactions at various levels. The geographical and epidemiological overlap increases risk for co-infection and co-treatment. The immune suppression due to HIV increases malaria incidence, severity and risk for poor treatment outcomes including mortality and adverse pregnancy outcomes such as anemia and low birth weight. Malaria infection increases HIV viral replication. Both malaria and HIV are treated with combination therapy to enhance treatment outcomes and reduce risk for development of resistance, consequently creating potential for drug-drug interactions (DDIs) when the two diseases are treated concomitantly. Previous studies demonstrated significant reduction in systemic exposure to Artemether, its metabolite dihydroartemisinin, and the long acting partner drug lumefantrine when the ACT artemether-lumefantrine was co-administered with efavirenz-based ART to HIV-malaria co-infected individuals.

Exposure to sub therapeutic antimalarial drug concentrations poses a risk for poor malaria treatment outcomes such as prolonged morbidity, anemia, death and poor birth outcomes for pregnant women plus increased economic costs and risk for drug resistance. There are currently limited drug options available for both malaria and HIV treatment especially in sub-Saharan Africa, thus the need to protect drug effectiveness. There are very scanty data on effects of drug interactions on malaria clinical outcomes, and such studies would be unethical currently. Despite these gaps, co-administration of antimalarial and antiretroviral drugs occurs with no guidance on therapeutic interventions to overcome these deleterious effects. Data are therefore urgently needed to optimize treatment of malaria for HIV-malaria co-infected individuals.

General Objective: To utilize innovative interventions to overcome drug interactions between artemether-lumefantrine and efavirenz to guide malaria treatment for individuals co-infected with HIV and malaria.

Specific objectives:

Objectives

1. To determine the safety and Pharmacokinetics of the double dose artemether-lumefantrine when administered to healthy volunteers (malaria negative and HIV negative individuals).
2. To determine the safety and Pharmacokinetics of the 5-day course of artemether-lumefantrine when administered to healthy volunteers (malaria negative and HIV negative individuals).
3. To determine the safety, pharmacokinetics and malaria treatment outcome of a standard dose of artemether-lumefantrine compared to double of the standard dose for weight and a 5-day course of artemether-lumefantrine for treatment of uncomplicated malaria among HIV-Malaria co-infected individuals receiving efavirenz (400mg) based ART.
4. To determine the safety and Pharmacokinetics of artemether-lumefantrine when administered with Dolutegravir based ART among HIV-malaria co-infected individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Willing and able to comply with study treatment and procedures
3. Age above 18 years
4. Confirmed HIV positive and receiving efavirenz or dolutegravir based ART for objectives 3 and 4
5. Confirmed Malaria blood film positive without evidence for severe malaria for objectives 3 and 4
6. Confirmed Malaria blood film negative for objectives 1 and 2

Exclusion Criteria:

1. Serum alanine transaminase levels above 3x upper limit of normal
2. Serum creatinine levels above 2x upper limit of normal
3. Use of known inducers/inhibitors of CYP or glucuronyl transferase UGT1A1 within past 2 months (e.g. anticonvulsants, TB medications, HIV agents for prophylaxis, azole antifungals)
4. Pregnant women or female subjects who are unwilling to use a suitable contraceptive method for the duration of the study (condom, diaphragm, IUD or contraceptive implant)
5. Likely to be poorly adherent based on clinician's medical judgement
6. Known to be current injection drug user
7. Administration of any additional antimalarial drugs that are not study drugs within 24 hours before study enrollment and during the course of the study.
8. Presence of any non-malarial febrile illness which may interfere with the classification of malaria treatment outcome
9. Movement away from the study area interfering with follow-up assessment
10. Patients with contraindications to taking the study drugs
11. Evidence of QT prolongation on ECG (rate adjusted QT interval>45ms (men (or >470ms for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 888 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Measure of malaria treatment outcome adjusted by genotyping and classified as reinfection or recrudescence. | Day 42
  The Primary outcome measure will be the malaria treatment outcome adjusted by genotyping and classified as reinfection or recrudescence.
  Treatment outcomes will be classified on the basis of an assessment of the parasitological and clinical outcomes of antimalarial treatment according to the latest WHO guidelines. Thus, all patients will be classified as having early treatment failure, late clinical failure, late parasitological failure or an adequate clinical and parasitological response.
  Clinical Treatment outcomes will be assessed according to WHO criteria as; early treatment failure and late treatment failure. Parasitological treatment outcomes will be classified as late parasitological failure and adequate clinical and parasitological response.

SECONDARY OUTCOMES:
Change Maximum concentration [Cmax] of the antimalarials (Artemether, dihydroartemisinin [DHA], lumefantrin and desbutylumefantrine | over 120hours
  Plots of plasma concentration versus time curves will be produced for artemether, dihydroartemisinin, lumefantrine and desbutyl-lumefantrine. Pharmacokinetic parameter Cmax derived directly from the data. The Cmax pharmacokinetic parameter will be presented using descriptive summary statistics including geometric means, geometric mean ratios (GMR) and confidence intervals (CI), or medians and interquartile ranges. The CIs will be determined using logarithms of the individual geometric mean values; the calculated values will be then expressed as linear values.
Measuring level of Hemoglobin | Hemoglobin will be measured from on follow-up days; 7, 14, 21 and 28.
  Anemia is a common with Malaria. The hemoglobin levels will be measured to assess for any reduction and also recovery of the hemoglobin level following treatment.
Change in Area under the time-concentration curve [AUC] of the antimalarials (Artemether, dihydroartemisinin [DHA], lumefantrin and desbutylumefantrine | over 120hours
  Plots of plasma concentration versus time curves will be produced for artemether. AUC over 24 hours (AUC0-24) will be calculated using non-compartmental methods (WinNonlin® Version 6.2, Pharsight). The pharmacokinetic parameter will be presented using descriptive summary statistics including geometric means, geometric mean ratios (GMR) and confidence intervals (CI), or medians and interquartile ranges. The CIs will be determined using logarithms of the individual geometric mean values; the calculated values will be then expressed as linear values.
Change in Time to maximum concentration [Tmax] of the antimalarials (Artemether, dihydroartemisinin [DHA], lumefantrin and desbutylumefantrine) | over 120hours
  Plots of plasma concentration versus time curves will be produced for artemether, dihydroartemisinin, lumefantrine and desbutyl-lumefantrine. Pharmacokinetic parameter time to maximal concentration (Tmax) will be derived directly from the data. The pharmacokinetic parameter will be presented using descriptive summary statistics including geometric means, geometric mean ratios (GMR) and confidence intervals (CI), or medians and interquartile ranges. The CIs will be determined using logarithms of the individual geometric mean values; the calculated values will be then expressed as linear values.
Change in Clearance [Cl/F] of the antimalarials (Artemether, dihydroartemisinin [DHA], lumefantrin and desbutylumefantrine) | over 120hours
  Plots of plasma concentration versus time curves will be produced for artemether, dihydroartemisinin, lumefantrine and desbutyl-lumefantrine. The apparent oral clearance will be calculated using non-compartmental methods (WinNonlin® Version 6.2, Pharsight). This pharmacokinetic parameter will be presented using descriptive summary statistics including geometric means, geometric mean ratios (GMR) and confidence intervals (CI), or medians and interquartile ranges. The CIs will be determined using logarithms of the individual geometric mean values; the calculated values will be then expressed as linear values.
Change in Trough concentration [Ctrough]) of the antimalarials (Artemether, dihydroartemisinin [DHA], lumefantrin and desbutylumefantrine) | over 120hours
  Plots of plasma concentration versus time curves will be produced for artemether, dihydroartemisinin, lumefantrine and desbutyl-lumefantrine. The change in trough concentration will be presented using descriptive summary statistics including geometric means, geometric mean ratios (GMR) and confidence intervals (CI), or medians and interquartile ranges. The CIs will be determined using logarithms of the individual geometric mean values; the calculated values will be then expressed as linear values.
Prolongation of the QT interval | Over 35days
  ECG Monitoring A 12-lead ECG to monitor for QT prolongation will be performed. If any prolongation of the QT interval is observed, the ECGs will be performed at every study visit until normalization.
Change in the level on the liver enzymes ALT and ALP | Over 35days
  Liver Function will be assessed at screening, and on days 7 and 35. Should any derangement in function be observed, the same will be performed at every study visit until normalization. Any participant with deranged liver function will be reported to have either adverse event or serious adverse event depending on the degree of severity and will be further assessed, treated appropriately and followed up till resolution
Change in creatinine and urea levels | Over 35days
  Renal Function will be assessed at screening, and on days 7 and 35. Should any derangement in function be observed, the same will be performed at every study visit until normalization. Any participant with deranged renal function (Creatinine and urea levels) will be reported to have either adverse event or serious adverse event depending on the degree of severity and will be further assessed, treated appropriately and followed up till resolution" Focus will be on monitoring change

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Byakika-Kibwika, PHD, Principal Investigator — IDI
Locations (2):
- Uganda (2):
  - Infectious Diseases Institute, Kampala
  - Tororo District Hospital, Tororo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF, CSR